CLINICAL TRIAL: NCT03935204
Title: An Randomized, Double-Blinded, Placebo Controlled Phase II Clinical Trial to Estimate Immunogenicity of the Recombinant Human Papillomavirus Vaccine (6,11,16,18,31,33,45,52,58 Type) (E.Coli) in Healthy Adults Aged 18 to 45 Years
Brief Title: Immunogenicity Study of Recombinant Human Papillomavirus Vaccine(6,11,16,18,31,33,45,52,58 Type)(E.Coli)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xiamen University (Other)
Collaborators: Xiamen Innovax Biotech Co., Ltd (Industry); Beijing Wantai Biological Pharmacy Enterprise Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jun Zhang, professor, Xiamen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HPV-PRO-008
Record Dates: First submitted 2019-04-30; First posted 2019-05-02 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Condylomata Acuminata; Cervical Cancer
Keywords: human papillomavirus vaccine
MeSH Terms: conditions — Condylomata Acuminata; Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HPV Vaccine,270μg/1.0ml (Experimental): Participants in this arm would receive 270μg/1.0ml HPV vaccines.
  Interventions: Biological: HPV Vaccine,270μg/1.0ml
- Placebo (Placebo Comparator): Participants in this arm would receive 1.0ml aluminium adjuvant.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: HPV Vaccine,270μg/1.0ml — HPV vaccine (270μg/1.0ml) administered intramuscularly according to a 0, 1, 6 month vaccination schedule.
  Arms: HPV Vaccine,270μg/1.0ml
Biological: Placebo — Aluminium adjuvant (1.0ml) administered intramuscularly according to a 0, 1, 6 month vaccination schedule.
  Other Names: aluminium adjuvant
  Arms: Placebo

SUMMARY:
This phase II clinical study was designed to evaluate the immunogenicity and safety of Recombinant Human Papillomavirus Vaccine (6,11,16,18,31,33,45,52,58 Type)(E.Coli)(hereafter called HPV vaccine), manufactured by Xiamen Innovax Biotech CO., LTD., in healthy adults aged 18-45 years old.

ELIGIBILITY:
Inclusion Criteria:

1. Health women aged between 18 and 45 years.
2. Judged as healthy and eligible for vaccination by the investigators through a self-reported medical history and some physical examinations.
3. Able to comply with the requests of the study.
4. Written informed consent obtained from the participants.
5. Axillary temperature not higher than 37.0°C
6. Non-pregnant women verified by a urine pregnancy test.

Exclusion Criteria:

1. Pregnant or breastfeeding or plan to be pregnant within 7 months.
2. Use of any investigational product or non-registered product (drug or vaccine) within 30 days preceding the first dose of the study vaccine or plan to use during the study period.
3. Received immunosuppressed, immunoregulation therapy or corticosteroid systemic therapy for more than 14 days in the 6 months before entry, except local treatment.
4. Administration of any immunoglobulin or blood products within 3 months preceding the first dose of the study vaccine or plan to use within 7 months.
5. Administration of any attenuated live vaccines within 21 days preceding the first dose of the study vaccine or any subunit or inactivated vaccines within 14 days before vaccination.
6. Had a fever (axillary temperature over 38°C) within 3 days or acute illness requiring systemic antibiotics or antiviral treatment within 5 days before vaccination.
7. Having the plan to participate another clinical trial during the study period.
8. Received another HPV vaccine.
9. Immunodeficiency , primary disease of important organs, malignant tumor, or any immune disease (such as systemic lupus erythematosus, arthritis pauperum, splenectomy or functional asplenia or other disease which might affect immune response).
10. History of allergic disease or history of serious adverse events occurring after vaccination, i.e., allergy, urticaria, dyspnea, angioneurotic edema or abdominal pain.
11. Asthma that required emergent treatment, hospitalization, oral or intravenous corticosteroid for unstable condition within the past 2 years.
12. Having serious disease of internal medicine, such as hypertension, cardiac disease, diabetes, hyperthyroidism et al.
13. Diagnosed coagulant function abnormality or blood coagulation disorder.
14. Epilepsy, except fever epilepsy at under 2 years of age, alcohol-induced epilepsy in 3 years before abstinence, or idiopathic epilepsy requiring no treatment in the past 3 years.
15. Past or current two-stage affective psychosis, not well controlled in the past 2 years or requiring drugs, or hve a tendency to commit suicide in the past 5 years.
16. Other medical, psychological, social or occupational factors that, according to the investigators' judgment, might affect the individual's ability to obey the protocol or sign the informed consent.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 627 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Anti-HPV 6, 11, 16, 18, 31, 33, 45, 52, and 58 seroconversion rates and geometric mean concentrations at Months 7 (type specific neutralizing antibody) | month 7
  To detect the anti-HPV 6, 11, 16, 18, 31, 33, 45, 52, and 58 type specific neutralizing antibody level on day 0 (before the 1st dose) and one month after dose 3

SECONDARY OUTCOMES:
Solicited local adverse reactions | During the 7-day (Day 0-6) period following each vaccination
  Solicited local adverse reactions occurred within 7 days after each vaccination;
Solicited systematic adverse reactions | During the 7-day (Day 0-6) period following each vaccination
  Solicited systematic adverse reactions occurred within 7 days after each vaccination;
Unsolicited adverse events | Within 30 days (Day 0-29) after any vaccination
  Unsolicited adverse reactions occurred within 30 days after each vaccination;
Serious adverse events | throughout the study period, an average of 7 months
  Serious adverse events occurred throughout the study;

OTHER OUTCOMES:
Anti-HPV 6, 11, 16, 18, 31, 33, 45, 52, and 58 seroconversion rates and geometric mean concentrations at Months 7 (type specific IgG antibody) | month 7
  To detect the anti-HPV 6, 11, 16, 18, 31, 33, 45, 52, and 58 type specific IgG antibody level on day 0 (before the 1st dose) and one month after dose 3
Anti-HPV 6, 11, 16, 18, 31, 33, 45, 52, and 58 seroconversion rates and geometric mean concentrations in a immunogenicity subgroup at Months 1,2 and 7 (type specific neutralizing antibody and IgG antibody) | month 1,2 and 6
  To detect the anti-HPV 6, 11, 16, 18, 31, 33, 45, 52, and 58 type specific neutralizing and IgG antibody level of a immunogenicity subgroup at month 1,2 and 6.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, Master, Study Chair — Xiamen University; Yue-Mei Hu, Bachelor, Principal Investigator — Jiangsu Provincial Centre for Disease Control and Prevention
Locations (1):
- Jiangsu Provincial Centre for Disease Control and Prevention, Nanjing, Jiangsu, China